CLINICAL TRIAL: NCT04529538
Title: A First-in-human, Phase 1, Randomized, Observer-blind, Controlled Study to Assess the Safety and Immunogenicity of Novel Live Attenuated Type 1 and Type 3 Oral Poliomyelitis Vaccines in Healthy Adults
Brief Title: Study of Novel Types 1 and 3 Oral Poliomyelitis Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); Viroclinics Biosciences B.V. (Industry); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CVIA 076
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Poliomyelitis
Keywords: Vaccine tolerability; Vaccine reactogenicity; Vaccine viral shedding; Vaccine immunogenicity
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Intervention Model Description: It will be an 8-arm, randomized, observer-blind, controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group1: nOPV1 (IPV History) (Experimental): Healthy adults fully vaccinated against polio exclusively by IPV were administered 1 vaccination of novel OPV type 1 (nOPV1) containing 10^6.5 cell culture infectious dose 50% (CCID50) on Day 1.
  Interventions: Biological: Novel Oral Polio Vaccine Type 1 (nOPV1)
- Group 2: mOPV1 (IPV History) (Active Comparator): Healthy adults fully vaccinated against polio exclusively by IPV were administered 1 vaccination of mOPV1 containing 10^6.0 CCID50 on Day 1.
  Interventions: Biological: Sabin Monovalent Oral Polio Vaccine Type 1 (mOPV1)
- Group 3: nOPV1 (OPV History) (Experimental): Healthy adults fully vaccinated against polio with an OPV-containing vaccine history were administered 2 vaccinations of nOPV1 containing 10^6.5 CCID50/dose, given 28 days apart.
  Interventions: Biological: Novel Oral Polio Vaccine Type 1 (nOPV1)
- Group 4: mOPV1 (OPV History) (Active Comparator): Healthy adults fully vaccinated against polio with an OPV-containing vaccine history were administered 2 doses of mOPV1 containing ≥ 10^6.0 CCID50/dose, given 28 days apart.
  Interventions: Biological: Sabin Monovalent Oral Polio Vaccine Type 1 (mOPV1)
- Group 5: nOPV3 (IPV History) (Experimental): Healthy adults fully vaccinated against polio exclusively by IPV were administered 1 vaccination of nOPV3 containing 10^6.5 CCID50 on Day 1.
  Interventions: Biological: Novel Oral Polio Vaccine Type 3 (nOPV3)
- Group 6: mOPV3 (IPV History) (Active Comparator): Healthy adults fully vaccinated against polio by exclusively IPV were administered 1 vaccination of mOPV3 containing ≥ 10^5.8 CCID50 on Day 1.
  Interventions: Biological: Sabin Monovalent Oral Polio Vaccine Type 3 (mOPV3)
- Group 7: nOPV3 (OPV History) (Experimental): Healthy adults fully vaccinated against polio with an OPV-containing vaccine history were administered 2 vaccinations of nOPV3 in a dose of 10^6.5 CCID50/dose, given 28 days apart.
  Interventions: Biological: Novel Oral Polio Vaccine Type 3 (nOPV3)
- Group 8: mOPV3 (OPV History) (Active Comparator): Healthy adults fully vaccinated against polio with an OPV-containing vaccine history were administered 2 vaccinations of mOPV3 containing ≥ 10^5.8 CCID50/dose, given 28 days apart.
  Interventions: Biological: Sabin Monovalent Oral Polio Vaccine Type 3 (mOPV3)

INTERVENTIONS:
Biological: Novel Oral Polio Vaccine Type 1 (nOPV1) — Each 0.1 mL (2 drops) dose of vaccine contains approximately 10^6.5 CCID50.
  Arms: Group 3: nOPV1 (OPV History); Group1: nOPV1 (IPV History)
Biological: Novel Oral Polio Vaccine Type 3 (nOPV3) — Each 0.1 mL (2 drops) dose of vaccine contains approximately 10^6.5 CCID50.
  Arms: Group 5: nOPV3 (IPV History); Group 7: nOPV3 (OPV History)
Biological: Sabin Monovalent Oral Polio Vaccine Type 1 (mOPV1) — The Sabin mOPV1 control vaccine contains ≥ 10^6.0 CCID50 per 0.1 mL (2 drops) dose.
  Arms: Group 2: mOPV1 (IPV History); Group 4: mOPV1 (OPV History)
Biological: Sabin Monovalent Oral Polio Vaccine Type 3 (mOPV3) — the Sabin mOPV3 control vaccine contains ≥ 10^5.8 CCID50 per 0.1 mL (2 drops) dose.
  Other Names: Sabin monovalent oral polio vaccine type 3
  Arms: Group 6: mOPV3 (IPV History); Group 8: mOPV3 (OPV History)

SUMMARY:
The purpose of this study is to assess the safety (primary objective), the ability to trigger the production of antibodies (immunogenicity; a secondary objective) and presence of vaccine virus in the stool (fecal shedding; a secondary objective) of two novel oral polio vaccines (nOPV), novel oral poliomyelitis vaccine type 1 (nOPV1) and novel oral poliomyelitis vaccine type 3 (nOPV3), as compared to Sabin strain monovalent oral poliomyelitis vaccine (mOPV) controls, in healthy adults.

DETAILED DESCRIPTION:
This multicenter trial is the first-in-human assessment of two novel oral polio vaccines for poliovirus type 1 and type 3. It will be a 4-cohort, 8-arm, randomized, observer-blind, controlled trial, with Sabin monovalent vaccines serving as the control for each type:

Cohort 1: Healthy adults with an exclusive inactivated poliovirus vaccine (IPV) prior vaccination history will be randomized in a 1:1 ratio and allocated to receive nOPV1 (Group 1) or mOPV1 (Group 2).

Cohort 2: Healthy adults with an OPV-containing prior vaccination history will be randomized in a 2:1 ratio and allocated to receive two doses of nOPV1 (Group 3) or mOPV1 (Group 4), respectively;

Cohort 3: Healthy adults with an exclusive IPV prior vaccination history will be randomized in a 1:1 ratio and allocated to receive nOPV3 (Group 5) or mOPV3 (Group 6);

Cohort 4: Healthy adults with an OPV-containing prior vaccination history will be randomized in a 2:1 ratio to study groups 3 and 4 and allocated to receive two doses of nOPV3 (Group 7) or mOPV3 (Group 8), respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, from 18 to 45 years of age (inclusive) at the time of enrollment
2. Healthy, as defined by the absence of any clinically significant medical conditions, either acute or chronic, as determined by medical history, physical examination, screening laboratory test results, and clinical assessment of the investigator
3. Willing and able to provide written informed consent prior to performance of any study-specific procedure
4. If female and of childbearing potential*, be not breastfeeding and not pregnant (based on a negative serum pregnancy test at screening and a negative urine pregnancy test during the 24 hours prior to any study vaccination), agreeing to have repeated pregnancy tests prior to any study vaccination, and having practiced adequate contraception** for 30 days prior to first study vaccination and willing to continue using adequate contraception consistently for at least 90 days after the last study vaccination and until cessation of vaccine virus shedding is confirmed

   * Females can be considered not of childbearing potential if they are with current bilateral tubal ligation, occlusion or removal, or post-total hysterectomy, or post-bilateral ovariectomy

   ** Adequate contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label, for example:
   * Abstinence from penile-vaginal intercourse
   * Combined estrogen and progesterone oral contraceptives
   * Hormonal (e.g., progestogen) injections
   * Hormonal (e.g., etonogestrel or levonorgestrel) implants
   * Contraceptive vaginal ring
   * Percutaneous contraceptive patches
   * Intrauterine device
   * Intrauterine hormonal system
   * Male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository), and/or progesterone alone oral contraceptive
   * Monogamous relationship with vasectomized (≥ 180 days prior to enrollment) partner
5. Resides in study area and is able and willing to adhere to all study restrictions and to all study visits and procedures (as evidenced by a signed informed consent form [ICF] and assessment by the investigator)
6. Agrees not to and has no plans to travel outside the United States (US) until confirmation of cessation of vaccine virus shedding in stool at or after the study Day 57 stool collection
7. Able and willing to be contacted by telephone or text, and willing for study staff to leave telephone voice or electronic messages as needed
8. Neutralizing antibody titer ≥ 1:8 for poliovirus type 1 (for participants in cohorts 1 and 2) and ≥ 1:8 for poliovirus type 3 (for participants in cohorts 3 and 4)
9. For Cohorts 1 and 3 only: previously received at least 3 doses of IPV and with no history of receipt of OPV. For Cohorts 2 and 4 only: previously received a primary polio immunization series containing OPV

Exclusion Criteria:

1. Have any condition (medical, psychiatric or behavioral) that, in the opinion of the investigator, would increase the participant's health risks in study participation or would increase the risk of not achieving the study's objectives (e.g., would compromise adherence to protocol requirements or interfere with planned safety and immunogenicity assessments)
2. Receipt of polio vaccine within 12 months before the start of the study
3. Having Crohn's disease or ulcerative colitis or having had major surgery of the gastrointestinal tract involving significant loss or resection of the bowel
4. A known allergy, hypersensitivity, or intolerance to any components of the study vaccines, including all macrolide and aminoglycoside antibiotics (e.g., erythromycin and kanamycin)
5. Any confirmed or suspected immunosuppressive or immunodeficiency condition (human immunodeficiency virus [HIV] infection, or total serum immunoglobulin A (IgA) or immunoglobulin G (IgG) level below the testing laboratory's lower limit of normal [LLN])
6. Administration of any long-acting immune-modifying drugs (e.g., infliximab or rituximab) or the chronic administration (i.e., longer than 14 days) of immunosuppressant drugs (e.g., oral or systemic steroids) or other immune-modifying drugs within 6 months prior to the first vaccine dose or planned use during the study (inhaled and topical steroids are allowed whereas intraarticular and epidural injection/administration of steroids are not allowed)
7. Will have household direct or close professional contact during the study with individuals expected to be immunosuppressed (due to underlying condition or treatments) or individuals who have not yet completed their primary infant polio immunization series (i.e., three doses)
8. Will have household direct or close professional contact during the study with pregnant women
9. Will have household direct or close professional (e.g., neonatal nurses) contact during the study with children less than 2 years of age or with individuals who are encopretic (i.e., infants/toddlers who are not yet toilet trained or other individuals, including adults, with fecal incontinence)
10. Will have professional handling of food, catering, or food production activities during the study
11. Reside in homes with septic tanks
12. Acute illness or fever (body temperature measured orally ≥ 38°C or 100.4°F) at the time of study vaccine administration (once acute illness/fever is resolved, if appropriate, as per investigator assessment, participant may complete screening)
13. Indications of drug abuse or excessive use of alcohol as deemed by the investigator to confound safety assessments or render the participant unable or unlikely to adhere to protocol requirements or provide accurate safety reports
14. Participation in another investigational product (drug or vaccine) clinical trial within 30 days prior to entry in this study or receipt of any such investigational product other than the study vaccine within 30 days prior to the first administration of study vaccine, or planned use during the study period
15. Administration of any vaccine (except seasonal inactivated influenza and COVID-19 vaccines which are prohibited for only 14 days prior to or following each study vaccination) other than the study vaccine or any intramuscular injection within 30 days prior to the first dose of study vaccine or planned administration within 30 days prior to or after any study vaccination.
16. Receipt of transfusion of any blood product or application of immunoglobulins within the 12 weeks prior to the first administration of study vaccine or planned use during the study period
17. Hepatitis B or C virus infection
18. Any hematological# or chemistry** parameter that is out of range of normal†† and is considered clinically significant by the investigator

    #Complete blood count (CBC), includes hemoglobin, hematocrit, white blood cell (WBC) count, neutrophil count, lymphocyte count, eosinophil count, and platelet count

    **Creatinine, alanine transaminase (ALT), total bilirubin

    ††Per the site clinical laboratory's reference ranges. All tests with out of range results that are regarded as clinically significant by the clinician must be repeated and determined to be not clinically significant before any participant can be enrolled.
19. The following hematological or chemistry laboratory results will be considered exclusionary, irrespective of assessment of clinical significance:

    * Hemoglobin (Male) < 12.5 g/dL
    * Hemoglobin (Female) < 11.0 g/dL
    * Neutrophil count < 1,000 cells/mm^3
    * Eosinophil count > 650 cells/mm^3
    * Platelet count < 125,000 cells/mm^3
    * Creatinine > 1.4 mg/dL
    * ALT > 1.1 X upper limit of normal (ULN) (per the site clinical laboratory's reference ranges)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Crothers, MD, Principal Investigator — University of Vermont; Arlene Sena, MD, Principal Investigator — University of North Carolina; Peter Wright, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Mohamed Al-Ibrahim, MB CHB, FACP, Principal Investigator — Pharmaron CPC, Inc.
Locations (4):
- United States (4):
  - Pharmaron CPC, Inc., Baltimore, Maryland
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of North Carolina Institute for Global Health and Infectious Diseases (IGHID), Chapel Hill, North Carolina
  - University of Vermont Vaccine Testing Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mercer LD, Sena AC, Colgate ER, Crothers JW, Wright PF, Al-Ibrahim M, Tritama E, Vincent A, Mainou BA, Zhang Y, Konopka-Anstadt J, Bandyopadhyay AS, Fix A, Konz JO, Gast C. Safety and immunogenicity of novel live attenuated type 1 and type 3 oral poliomyelitis vaccines in healthy adults in the USA: a first-in-human, observer-masked, multicentre, phase 1 randomised controlled trial. Lancet Infect Dis. 2025 Dec;25(12):1363-1376. doi: 10.1016/S1473-3099(25)00285-3. Epub 2025 Aug 13. PMID 40818478
- [Derived] Thompson KM, Kalkowska DA, Kidd SE, Burns CC, Badizadegan K. Trade-offs of different poliovirus vaccine options for outbreak response in the United States and other countries that only use inactivated poliovirus vaccine (IPV) in routine immunization. Vaccine. 2024 Feb 6;42(4):819-827. doi: 10.1016/j.vaccine.2023.12.081. Epub 2024 Jan 12. PMID 38218668

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were enrolled at four study sites in the United States. This study consisted of 4 cohorts, each with 2 groups of participants.
  Participants must have received either prior vaccination with at least 3 doses of inactivated poliovirus vaccine (IPV) with no history of receipt of oral poliomyelitis vaccine (OPV) (Cohorts 1 and 3) or previously received a primary polio immunization series containing OPV (Cohorts 2 and 4).
Pre-assignment Details: Cohorts 1 and 2 received vaccine against poliovirus type 1 and Cohorts 3 and 4 received vaccine against poliovirus type 3.
  In Cohorts 1 and 3 participants with an exclusive IPV vaccination history were randomized in a 1:1 ratio to receive novel oral poliomyelitis vaccine (nOPV) or Sabin strain monovalent oral poliomyelitis vaccine (mOPV) control.
  In Cohorts 2 and 4, participants with an OPV-containing vaccination history were randomized in a 2:1 ratio to receive nOPV or mOPV.
Groups:
- Group1: nOPV1 (IPV History): Healthy adults fully vaccinated against polio exclusively by IPV were administered 1 vaccination of novel oral polio vaccine type 1 (nOPV1) containing 10^6.5 cell culture infectious dose 50% (CCID50) on Day 1.
- Group 2: mOPV1 (IPV History): Healthy adults fully vaccinated against polio exclusively by IPV were administered 1 vaccination of Sabin monovalent oral polio vaccine type 1 (mOPV1) containing 10^6.0 CCID50 on Day 1.
- Group 4: mOPV1 (OPV History): Healthy adults fully vaccinated against polio with an OPV-containing vaccine history were administered 2 doses of Sabin mOPV1 containing ≥ 10^6.0 CCID50/dose, given 28 days apart.
- Group 5: nOPV3 (IPV History): Healthy adults fully vaccinated against polio exclusively by IPV were administered 1 vaccination of novel oral poliomyelitis vaccine type 3 (nOPV3) containing 10^6.5 CCID50 on Day 1.
- Group 6: mOPV3 (IPV History): Healthy adults fully vaccinated against polio by exclusively IPV were administered 1 vaccination of Sabin monovalent oral polio vaccine type 3 (mOPV3) containing ≥ 10^5.8 CCID50 on Day 1.
- Group 7: nOPV3 (OPV History): Healthy adults fully vaccinated against polio with an OPV-containing vaccine history were administered 2 vaccinations of nOPV3 containing 10^6.5 CCID50/dose, given 28 days apart.
Period: Overall Study
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History) | Group 3: nOPV1 (OPV History) | Group 4: mOPV1 (OPV History) | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History) | Group 7: nOPV3 (OPV History) | Group 8: mOPV3 (OPV History)
Started | 21 | 23 | 53 | 27 | 20 | 21 | 40 | 21
Received 1st Vaccination | 20 | 20 | 50 | 25 | 19 | 17 | 35 | 19
Received 2nd Vaccination | 0 (Not applicable as participants previously vaccinated with IPV only received 1 vaccination in this study) | 0 (Not applicable as participants previously vaccinated with IPV only received 1 vaccination in this study) | 49 | 22 | 0 (Not applicable as participants previously vaccinated with IPV only received 1 vaccination in this study) | 0 (Not applicable as participants previously vaccinated with IPV only received 1 vaccination in this study) | 35 | 18
Completed | 18 | 18 | 49 | 22 | 19 | 17 | 35 | 19
Not Completed | 3 | 5 | 4 | 5 | 1 | 4 | 5 | 2
Not completed — Lost to Follow-up | 3 | 2 | 1 | 0 | 1 | 1 | 2 | 0
Not completed — Not eligible at enrollment | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2 | 0 | 2 | 3 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population was defined as all participants who provided informed consent and who received a study vaccine, and for whom no potential transmission events between participants were identified by next generation sequencing of shed virus (Cohorts 1 and 3 only).
Groups:
- Group1: nOPV1 (IPV History): Healthy adults fully vaccinated against polio exclusively by IPV were administered 1 vaccination of nOPV1 containing 10^6.5 CCID50 on Day 1.
- Group 2: mOPV1 (IPV History): Healthy adults fully vaccinated against polio exclusively by IPV were administered 1 vaccination of Sabin mOPV1 containing 10^6.0 CCID50 on Day 1.
- Group 6: mOPV3 (IPV History): Healthy adults fully vaccinated against polio by exclusively IPV were administered 1 vaccination of Sabin mOPV3 containing ≥ 10^5.8 CCID50 on Day 1.
- Total: Total of all reporting groups
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History) | Group 3: nOPV1 (OPV History) | Group 4: mOPV1 (OPV History) | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History) | Group 7: nOPV3 (OPV History) | Group 8: mOPV3 (OPV History) | Total
Number analyzed (Participants) | 18 | 18 | 50 | 25 | 19 | 15 | 35 | 19 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (2.6) | 20.0 (1.6) | 30.0 (6.3) | 30.0 (6.5) | 20.7 (2.1) | 21.5 (2.4) | 30.4 (6.6) | 33.1 (8.8) | 27.1 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 25 | 15 | 10 | 7 | 21 | 13 | 110
  Male | 8 | 9 | 25 | 10 | 9 | 8 | 14 | 6 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 6 | 0 | 2 | 0 | 2 | 0 | 10
  Not Hispanic or Latino | 18 | 18 | 44 | 24 | 17 | 13 | 33 | 19 | 186
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 5 | 1 | 1 | 1 | 3 | 1 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 1 | 5 | 2 | 17 | 9 | 38
  White | 16 | 16 | 40 | 22 | 13 | 9 | 12 | 8 | 136
  More than one race | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event is any adverse event that resulted in any of the following outcomes:
  * Death
  * Was life-threatening
  * Required inpatient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * Congenital anomaly or birth defect
  * Important medical event that may not result in one of the above outcomes but may jeopardize the health of the study participant and/or require medical or surgical intervention to prevent one of the outcomes listed above
Time Frame: From Day 1 to end of study, up to 169 days
Population: The Reactogenicity Population was defined as all participants who provided informed consent and received a study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History) | Group 3: nOPV1 (OPV History) | Group 4: mOPV1 (OPV History) | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History) | Group 7: nOPV3 (OPV History) | Group 8: mOPV3 (OPV History)
Number analyzed (Participants) | 20 | 20 | 50 | 25 | 19 | 17 | 35 | 19
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited Adverse Events (AEs) 7 Days After First Dose of Study Vaccine
Description: Solicited AEs are pre-specified AEs that are common or known to be associated with vaccination that are actively monitored as potential indicators of vaccine reactogenicity. Solicited AEs for this study included:
  * Fever (oral temperature ≥ 38.0°C or 100.4°F)
  * Chills
  * Fatigue
  * Headache
  * Muscle aches/myalgias
  * Joint aches/arthralgias
  * Nausea
  * Vomiting
  * Abdominal pain
  * Diarrhea
Time Frame: From vaccination to 7 days post vaccination (Days 1-7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History) | Group 3: nOPV1 (OPV History) | Group 4: mOPV1 (OPV History) | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History) | Group 7: nOPV3 (OPV History) | Group 8: mOPV3 (OPV History)
Number analyzed (Participants) | 20 | 20 | 50 | 25 | 19 | 17 | 35 | 19
Participants
  Any Solicited Event | 11 | 12 | 25 | 15 | 10 | 9 | 13 | 7
  Fever | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills | 1 | 5 | 1 | 1 | 1 | 0 | 1 | 0
  Fatigue | 5 | 8 | 17 | 9 | 7 | 7 | 9 | 5
  Headache | 5 | 7 | 10 | 7 | 3 | 5 | 6 | 3
  Muscle Aches/Myalgias | 2 | 6 | 6 | 3 | 2 | 2 | 1 | 2
  Joint Aches/Arthralgias | 1 | 4 | 2 | 2 | 1 | 2 | 1 | 1
  Nausea | 2 | 2 | 6 | 2 | 1 | 1 | 8 | 0
  Vomiting | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
  Abdominal pain | 5 | 5 | 4 | 3 | 6 | 1 | 5 | 2
  Diarrhea | 2 | 4 | 9 | 6 | 3 | 6 | 3 | 3

3. Primary Outcome: Number of Participants With Solicited Adverse Events 7 Days After Second Dose of Study Vaccine
Description: as for outcome 2
Time Frame: From Day 29 to Day 35
Population: The Reactogenicity Population was defined as all participants who provided informed consent and received a study vaccine. The analysis includes groups / participants who received a 2nd vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History) | Group 3: nOPV1 (OPV History) | Group 4: mOPV1 (OPV History) | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History) | Group 7: nOPV3 (OPV History) | Group 8: mOPV3 (OPV History)
Number analyzed (Participants) | 0 | 0 | 49 | 22 | 0 | 0 | 35 | 18
Participants
  Any Solicited Event |  |  | 16 | 12 |  |  | 6 | 7
  Fever |  |  | 1 | 0 |  |  | 0 | 1
  Chills |  |  | 1 | 2 |  |  | 0 | 1
  Fatigue |  |  | 8 | 6 |  |  | 1 | 3
  Headache |  |  | 9 | 5 |  |  | 3 | 2
  Muscle Aches/Myalgias |  |  | 4 | 3 |  |  | 1 | 1
  Joint Aches/Arthralgias |  |  | 1 | 4 |  |  | 1 | 0
  Nausea |  |  | 3 | 2 |  |  | 3 | 1
  Vomiting |  |  | 0 | 1 |  |  | 1 | 0
  Abdominal pain |  |  | 4 | 2 |  |  | 1 | 0
  Diarrhea |  |  | 4 | 4 |  |  | 3 | 3

4. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs) up to 28 Days Post Vaccination
Description: Unsolicited AEs are any AEs reported spontaneously by the participant, observed by the study personnel during study visits or those identified during review of medical records or source documents.
  In the absence of a diagnosis, abnormal physical examination findings or abnormal clinical safety laboratory test results that are assessed by the investigator to be clinically significant were reported as an AE.
Time Frame: From vaccination to 28 days post vaccination (Day 1-28 for 1st vaccination and Day 29-56 for the 2nd vaccination)
Population: Reactogenicity population; the analysis includes participants who received each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History) | Group 3: nOPV1 (OPV History) | Group 4: mOPV1 (OPV History) | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History) | Group 7: nOPV3 (OPV History) | Group 8: mOPV3 (OPV History)
Number analyzed (Participants) | 20 | 20 | 50 | 25 | 19 | 17 | 35 | 19
Participants
  After 1st dose | 7 | 7 | 21 | 10 | 4 | 1 | 3 | 2
  After 2nd dose: number analyzed (Participants) | 0 | 0 | 49 | 22 | 0 | 0 | 35 | 18
  After 2nd dose |  |  | 16 | 7 |  |  | 2 | 3

5. Secondary Outcome: Median Anti-poliovirus Type 1 Serum Neutralizing Antibody Titers at Baseline and Post-vaccination Among Participants With a Vaccine History of IPV
Description: Blood samples collected from participants for type-specific poliovirus neutralizing antibodies were analyzed at the Polio and Picornavirus Laboratory Branch at the United States Centers for Disease Control and Prevention (CDC).
  For all immunogenicity endpoints, data are presented separately by:
  * Prior vaccination history (exclusively IPV vs OPV), and
  * Type-specific poliovirus vaccine received (type 1 vs type 3).
Time Frame: Baseline and Day 29 (28 days post-vaccination)
Population: The Per-Protocol Population (PPP) for immunogenicity was defined as all participants in the Reactogenicity Population who provided a baseline and at least 1 post-vaccination evaluable serum sample and who received correct study vaccinations per randomization with no major protocol deviations that might interfere with the immunogenicity result. The PPP was determined separately for each time point.
  The analysis includes groups with prior IPV history who received vaccination with a type 1 OPV.
Measure: Median (95% Confidence Interval); unit: log₂ titer
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History)
Number analyzed (Participants) | 18 | 15
log₂ titer
  Baseline | 5.67 [5.34 to 7.33] | 6.00 [5.83 to 7.50]
  Day 29 | NA [NA to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂) | NA [NA to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂)

6. Secondary Outcome: Median Anti-poliovirus Type 1 Serum Neutralizing Antibody Titers at Baseline and Post-vaccination Among Participants With a Vaccine History of OPV
Time Frame: Baseline, Day 29 (28 days post-vaccination) and Day 57 (28 days after 2nd vaccination)
Population: The Per-Protocol Population (PPP) for immunogenicity was defined as all participants in the Reactogenicity Population who provided a baseline and at least 1 post-vaccination evaluable serum sample and who received correct study vaccinations per randomization with no major protocol deviations that might interfere with the immunogenicity result. The PPP was determined separately for each time point.
  The analysis includes groups with prior OPV history who received vaccination with a type 1 OPV.
Measure: Median (95% Confidence Interval); unit: log₂ titer
Arm/Group | Group 3: nOPV1 (OPV History) | Group 4: mOPV1 (OPV History)
Number analyzed (Participants) | 48 | 23
log₂ titer
  Baseline | 6.83 [6.17 to 7.83] | 7.17 [5.50 to 8.17]
  Day 29 | NA [NA to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂) | NA [10.17 to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂)
  Day 57: number analyzed (Participants) | 47 | 22
  Day 57 | NA [NA to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂) | NA [NA to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂)

7. Secondary Outcome: Median Anti-poliovirus Type 3 Serum Neutralizing Antibody Titers at Baseline and Post-vaccination Among Participants With a Vaccine History of IPV
Time Frame: Baseline and Day 29 (28 days post-vaccination)
Population: The Per-Protocol Population (PPP) for immunogenicity was defined as all participants in the Reactogenicity Population who provided a baseline and at least 1 post-vaccination evaluable serum sample and who received correct study vaccinations per randomization with no major protocol deviations that might interfere with the immunogenicity result. The PPP was determined separately for each time point.
  The analysis includes groups with prior IPV history who received vaccination with a type 3 OPV.
Measure: Median (95% Confidence Interval); unit: log₂ titer
Arm/Group | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History)
Number analyzed (Participants) | 19 | 15
log₂ titer
  Baseline | 6.17 [5.83 to 8.17] | 6.17 [5.50 to 6.83]
  Day 29 | NA [NA to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂) | NA [9.50 to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂)

8. Secondary Outcome: Median Anti-poliovirus Type 3 Serum Neutralizing Antibody Titers at Baseline and Post-vaccination Among Participants With a Vaccine History of OPV
Time Frame: Baseline, Day 29 (28 days after the 1st vaccination) and Day 57 (28 days after 2nd vaccination)
Population: The Per-Protocol Population (PPP) for immunogenicity was defined as all participants in the Reactogenicity Population who provided a baseline and at least 1 post-vaccination evaluable serum sample and who received correct study vaccinations per randomization with no major protocol deviations that might interfere with the immunogenicity result. The PPP was determined separately for each time point.
  The analysis includes groups with prior OPV history who received vaccination with a type 3 OPV.
Measure: Median (95% Confidence Interval); unit: log₂ titer
Arm/Group | Group 7: nOPV3 (OPV History) | Group 8: mOPV3 (OPV History)
Number analyzed (Participants) | 35 | 19
log₂ titer
  Baseline | 5.83 [4.17 to 6.83] | 6.50 [5.17 to 8.50]
  Day 29: number analyzed (Participants) | 34 | 19
  Day 29 | NA [NA to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂) | NA [9.50 to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂)
  Day 57: number analyzed (Participants) | 34 | 17
  Day 57 | NA [NA to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂) | 9.83 [9.17 to NA] — Titers above upper limit of quantitation (ULOQ) (10.5 log₂)

9. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-poliovirus Type 1 Serum Neutralizing Antibodies at Baseline and Post-vaccination Among Participants With a Vaccine History of IPV
Description: GMT and 95% confidence intervals are maximum likelihood estimates incorporating left and right censoring at the lower limit of quantitation (LLOQ) and ULOQ, respectively.
Time Frame: Baseline and Day 29 (28 days post-vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History)
Number analyzed (Participants) | 18 | 15
titer
  Baseline | 49.6 [26.7 to 92.1] | 73.2 [33.6 to 159.7]
  Day 29 | 5208.2 [904.6 to 29986.4] | 2846.7 [716.6 to 11307.6]
Statistical Analysis 1: Comparison: Group1: nOPV1 (IPV History) vs Group 2: mOPV1 (IPV History); Comparison of Type 1 neutralizing antibody GMT at Day 29; Test type: Other; GMT Ratio = 0.68, 95% CI 2-sided [0.252 to 1.838] — GMT ratios (nOPV/mOPV) were estimated via a linear model of the log₂ neutralizing antibody titer as a function of group with a fixed parameter for site and a covariate for the baseline log₂ neutralizing antibody titer level

10. Secondary Outcome: Geometric Mean Titer of Anti-poliovirus Type 1 Serum Neutralizing Antibodies at Baseline and Post-vaccination Among Participants With a Vaccine History of OPV
Time Frame: Baseline, Day 29 (28 days after 1st vaccination) and Day 57 (28 days after 2nd vaccination)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 3: nOPV1 (OPV History) | Group 4: mOPV1 (OPV History)
Number analyzed (Participants) | 48 | 23
titer
  Baseline | 111.6 [70.5 to 176.5] | 116.0 [48.1 to 280.1]
  Day 29 | 10869.2 [1953.5 to 60474.3] | 4495.1 [960.9 to 21027.0]
  Day 57: number analyzed (Participants) | 47 | 22
  Day 57 | 4407.5 [1547.8 to 12551.0] | 16500.8 [808.4 to 336813.5]
Statistical Analysis 1: Comparison: Group 3: nOPV1 (OPV History) vs Group 4: mOPV1 (OPV History); Comparison of type 1 neutralizing antibody GMT at Day 29; Test type: Other; GMT Ratio = 1.26, 95% CI 2-sided [0.232 to 6.833] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Group 3: nOPV1 (OPV History) vs Group 4: mOPV1 (OPV History); Comparison of type 1 neutralizing antibody GMT at Day 57; Test type: Other; GMT Ratio = 1.98, 95% CI 2-sided [0.603 to 6.528] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Geometric Mean Titer of Anti-poliovirus Type 3 Serum Neutralizing Antibodies at Baseline and Post-vaccination Among Participants With a Vaccine History of IPV
Time Frame: Baseline and Day 29 (28 days post-vaccination)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History)
Number analyzed (Participants) | 19 | 15
titer
  Baseline | 113.0 [56.7 to 225.2] | 74.6 [43.2 to 128.8]
  Day 29 | 3091.2 [1095.6 to 8721.9] | 3945.5 [736.6 to 21132.6]
Statistical Analysis 1: Comparison: Group 5: nOPV3 (IPV History) vs Group 6: mOPV3 (IPV History); Comparison of type 3 neutralizing antibody GMT at Day 29; Test type: Other; GMT Ratio = 1.56, 95% CI 2-sided [0.639 to 3.828] — [estimate comment as in outcome 9, analysis 1]

12. Secondary Outcome: Geometric Mean Titer of Anti-poliovirus Type 3 Serum Neutralizing Antibodies at Baseline and Post-vaccination Among Participants With a Vaccine History of OPV
Time Frame: Baseline, Day 29 (28 days after 1st vaccination) and Day 57 (28 days after 2nd vaccination)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 7: nOPV3 (OPV History) | Group 8: mOPV3 (OPV History)
Number analyzed (Participants) | 35 | 19
titer
  Baseline | 53.4 [29.1 to 97.8] | 101.1 [47.7 to 214.5]
  Day 29: number analyzed (Participants) | 34 | 19
  Day 29 | 2810.1 [1364.0 to 5789.3] | 1483.8 [758.8 to 2901.4]
  Day 57: number analyzed (Participants) | 34 | 17
  Day 57 | 3337.0 [1293.1 to 8611.7] | 1076.8 [613.5 to 1890.0]
Statistical Analysis 1: Comparison: Group 7: nOPV3 (OPV History) vs Group 8: mOPV3 (OPV History); Comparison of type 3 neutralizing antibody GMT at Day 29; Test type: Other; GMT Ratio = 1.79, 95% CI 2-sided [0.772 to 4.163] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Group 7: nOPV3 (OPV History) vs Group 8: mOPV3 (OPV History); Comparison of type 3 neutralizing antibody GMT at Day 57; Test type: Other; GMT Ratio = 2.51, 95% CI 2-sided [0.994 to 6.340] — [estimate comment as in outcome 9, analysis 1]

13. Secondary Outcome: Percentage of Participants With Any-Fold Rise, 2-fold Rise and 4-fold Rise in Anti-poliovirus Type 1 Serum Neutralizing Antibody Titers From Baseline to 28 Days After Vaccination Among Participants With a Vaccine History of IPV
Description: * Seroconversion (SCR) is defined as a minimum 4-fold increase in titer from Baseline (pre-vaccination) to 28 days post-vaccination among those participants with a 4-fold increase possible to observe, i.e., with a Baseline titer not greater than 8.5 log₂.
  * Minimum 2-fold-rise from Baseline to 28 days post-vaccination among those participants with a 2-fold increase possible to observe, i.e., with a Baseline titer not greater than 9.5 log₂.
  * Any fold-rise is defined as any increase in titer from Baseline to 28 days post-vaccination (log₂ neutralizing antibody titer post-dose minus Baseline > 0), among those with an increase possible to observe, i.e., with a Baseline titer less than 10.5 log₂.
Time Frame: Baseline (pre-vaccination) and Day 29 (28 days post-vaccination)
Population: Per Protocol Population. The analysis includes groups with prior IPV history who received vaccination with a type 1 OPV; participants were only included in each analysis if the appropriate measure could be observed based on Baseline neutralizing antibody titer.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History)
Number analyzed (Participants) | 18 | 14
percentage of participants
  ≥ 4-fold rise | 88.9 [65.29 to 98.62] | 92.9 [66.13 to 99.82]
  ≥ 2-fold rise | 94.4 [72.71 to 99.86] | 100 [76.84 to 100]
  Any fold-rise | 100 [81.47 to 100] | 100 [76.84 to 100]
Statistical Analysis 1: Comparison: Group1: nOPV1 (IPV History) vs Group 2: mOPV1 (IPV History); Between-Group Seroconversion Rate (4-fold rise) in Neutralizing Antibody Titers; Test type: Other; p > 0.999, Fisher Exact; Rate Difference = -4.0, 95% CI 2-sided [-27.67 to 22.72] — Rate Difference = nOPV - mOPV

14. Secondary Outcome: Percentage of Participants With Any-Fold Rise, 2-fold Rise and 4-fold Rise in Anti-poliovirus Type 1 Serum Neutralizing Antibody Titers From Baseline to 28 Days After Each Vaccination Among Participants With a Vaccine History of OPV
Description: as for outcome 13
Time Frame: Baseline, Day 29 (28 days post-vaccination) and Day 57 (28 days after 2nd vaccination)
Population: Per Protocol Population; The analysis includes groups with prior OPV history who received vaccination with a type 1 OPV; participants were only included in each analysis if the appropriate measure could be observed based on Baseline neutralizing antibody titer.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 3: nOPV1 (OPV History) | Group 4: mOPV1 (OPV History)
Number analyzed (Participants) | 47 | 20
percentage of participants
  Day 29: ≥ 4-fold rise: number analyzed (Participants) | 36 | 18
  Day 29: ≥ 4-fold rise | 86.1 [70.50 to 95.33] | 88.9 [65.29 to 98.62]
  Day 29: ≥ 2-fold rise: number analyzed (Participants) | 42 | 20
  Day 29: ≥ 2-fold rise | 83.3 [68.64 to 93.03] | 90.0 [68.30 to 98.77]
  Day 29: Any fold-rise | 83.0 [69.19 to 92.35] | 100 [83.16 to 100]
  Day 57: ≥ 4-fold rise: number analyzed (Participants) | 35 | 18
  Day 57: ≥ 4-fold rise | 97.1 [85.08 to 99.93] | 88.9 [65.29 to 98.62]
  Day 57: ≥ 2-fold rise: number analyzed (Participants) | 41 | 19
  Day 57: ≥ 2-fold rise | 95.1 [83.47 to 99.40] | 94.7 [73.97 to 99.87]
  Day 57: Any fold-rise: number analyzed (Participants) | 46 | 19
  Day 57: Any fold-rise | 97.8 [88.47 to 99.94] | 94.7 [73.97 to 99.87]
Statistical Analysis 1: Comparison: Group 3: nOPV1 (OPV History) vs Group 4: mOPV1 (OPV History); Between-group seroconversion rate (4-fold rise) in neutralizing antibody titers 28 days after first dose; Test type: Other; p > 0.999, Fisher Exact; Rate Difference = -2.8, 95% CI 2-sided [-20.47 to 20.86] — Rate Difference = nOPV - mOPV
Statistical Analysis 2: Comparison: Group 3: nOPV1 (OPV History) vs Group 4: mOPV1 (OPV History); Between-group comparison of seroconversion rate (4-fold rise) in neutralizing antibody titers 28 days after 2nd dose; Test type: Other; p = 0.263, Fisher Exact; Rate Difference = 8.3, 95% CI 2-sided [-5.71 to 30.57] — Rate Difference = nOPV - mOPV

15. Secondary Outcome: Percentage of Participants With Any-Fold Rise, 2-fold Rise and 4-fold Rise in Anti-poliovirus Type 3 Serum Neutralizing Antibody Titers From Baseline to 28 Days After Vaccination Among Participants With a Vaccine History of IPV
Description: as for outcome 13
Time Frame: Baseline and Day 29 (28 days post-vaccination)
Population: Per Protocol Population. The analysis includes groups with prior IPV history who received vaccination with a type 3 OPV; participants were only included in each analysis if the appropriate measure could be observed based on Baseline neutralizing antibody titer.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History)
Number analyzed (Participants) | 18 | 15
percentage of participants
  ≥ 4-fold rise: number analyzed (Participants) | 15 | 14
  ≥ 4-fold rise | 100 [78.20 to 100] | 85.7 [57.9 to 98.22]
  ≥ 2-fold rise: number analyzed (Participants) | 17 | 15
  ≥ 2-fold rise | 94.1 [71.31 to 99.85] | 100 [78.20 to 100]
  Any fold-rise | 94.4 [72.71 to 99.86] | 100 [78.20 to 100]
Statistical Analysis 1: Comparison: Group 5: nOPV3 (IPV History) vs Group 6: mOPV3 (IPV History); Between-group seroconversion rate (4-fold rise) in neutralizing antibody titers 28 days after vaccination; Test type: Other; p = 0.224, Fisher Exact; Rate Difference = 14.3, 95% CI 2-sided [-8.30 to 40.45] — Rate Difference = nOPV - mOPV

16. Secondary Outcome: Percentage of Participants With Any-Fold Rise, 2-fold Rise and 4-fold Rise in Anti-poliovirus Type 3 Serum Neutralizing Antibody Titers From Baseline to 28 Days After Each Vaccination Among Participants With a Vaccine History of OPV
Description: as for outcome 13
Time Frame: Baseline, Day 29 (28 days after 1st vaccination) and Day 57 (28 days after 2nd vaccination)
Population: Per Protocol Population; The analysis includes groups with prior OPV history who received vaccination with a type 3 OPV; participants were only included in each analysis if the appropriate measure could be observed based on Baseline neutralizing antibody titer.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 7: nOPV3 (OPV History) | Group 8: mOPV3 (OPV History)
Number analyzed (Participants) | 34 | 18
percentage of participants
  Day 29: ≥ 4-fold rise: number analyzed (Participants) | 28 | 15
  Day 29: ≥ 4-fold rise | 96.4 [81.65 to 99.91] | 86.7 [59.54 to 98.34]
  Day 29: ≥ 2-fold rise: number analyzed (Participants) | 32 | 18
  Day 29: ≥ 2-fold rise | 96.9 [83.78 to 99.92] | 83.3 [58.58 to 96.42]
  Day 29: Any fold-rise | 94.1 [80.32 to 99.28] | 94.4 [72.71 to 99.86]
  Day 57: ≥ 4-fold rise: number analyzed (Participants) | 28 | 14
  Day 57: ≥ 4-fold rise | 96.4 [81.65 to 99.91] | 78.6 [49.20 to 95.34]
  Day 57: ≥ 2-fold rise: number analyzed (Participants) | 34 | 17
  Day 57: ≥ 2-fold rise | 90.6 [74.98 to 98.02] | 76.5 [50.10 to 93.19]
  Day 57: Any fold-rise: number analyzed (Participants) | 32 | 17
  Day 57: Any fold-rise | 100 [89.72 to 100] | 88.2 [63.56 to 98.54]
Statistical Analysis 1: Comparison: Group 7: nOPV3 (OPV History) vs Group 8: mOPV3 (OPV History); Between-group comparison of seroconversion rate (4-fold rise) in neutralizing antibody titers 28 days after first dose; Test type: Other; p = 0.275, Fisher Exact; Rate Difference = 9.8, 95% CI 2-sided [-7.29 to 35.19] — Rate Difference = nOPV - mOPV
Statistical Analysis 2: Comparison: Group 7: nOPV3 (OPV History) vs Group 8: mOPV3 (OPV History); Between-group comparison of seroconversion rate (4-fold rise) in neutralizing antibody titers 28 days after 2nd dose; Test type: Other; p = 0.100, Fisher Exact; Rate Difference = 17.9, 95% CI 2-sided [-1.27 to 44.93] — Rate Difference = nOPV - mOPV

17. Secondary Outcome: Time to Cessation of Fecal Shedding of Vaccine Virus in Participants With IPV Vaccination History
Description: The presence of the vaccine virus in stool samples was assessed using polymerase chain reaction (PCR). Time to cessation of shedding is defined as the time between vaccination and the last PCR-positive stool prior to 2 consecutive PCR-negative stools (with a minimum 24-hour interval between the 2 negative stools). The time to cessation of fecal shedding of nOPV1 and nOPV3 in prior IPV recipients was estimated using Kaplan-Meier methodology with interval-censoring.
Time Frame: Up to Day 57
Population: Participants in the Safety Population with available PCR data; the analysis includes groups with prior IPV history.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History) | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History)
Number analyzed (Participants) | 18 | 18 | 19 | 15
days | 22 [15 to 24] | 20 [20 to 29] | 20 [15 to 37] | 29 [22 to 42]

18. Secondary Outcome: Time to Cessation of Fecal Shedding of Vaccine Virus in Participants With OPV Vaccination History
Description: The presence of the vaccine virus in stool samples was assessed using polymerase chain reaction (PCR). Time to cessation of shedding is defined as the time between vaccination and the last PCR-positive stool prior to 2 consecutive PCR-negative stools (with a minimum 24-hour interval between the 2 negative stools). The time to cessation of fecal shedding of nOPV1 and nOPV3 in prior OPV recipients was evaluated separately after each dose, estimated using Kaplan-Meier methodology with interval-censoring.
Time Frame: From vaccination through 28 days after each vaccination
Population: Participants in the Safety Population with available PCR data at each time point; the analysis includes groups with prior OPV history.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Group 3: nOPV1 (OPV History) | Group 4: mOPV1 (OPV History) | Group 7: nOPV3 (OPV History) | Group 8: mOPV3 (OPV History)
Number analyzed (Participants) | 50 | 25 | 35 | 19
days
  After first dose | 20 [9 to 20] | 20 [14 to 20] | 21 [13 to NA] — Could not be calculated due to low numbers of participants with positive shedding results | 17 [8 to NA] — Could not be calculated due to low numbers of participants with positive shedding results
  After 2nd dose: number analyzed (Participants) | 49 | 22 | 35 | 18
  After 2nd dose | 5 [NA to NA] — Could not be calculated due to low numbers of participants with positive shedding results | 7 [4 to 7] | 2 [NA to NA] — Could not be calculated due to low numbers of participants with positive shedding results | 2 [NA to NA] — Could not be calculated due to low numbers of participants with positive shedding results

19. Secondary Outcome: Percentage of Participants Shedding Type 1 Vaccine Virus at Each Post-vaccination Stool Collection in Participants With IPV Vaccination History
Description: Presence of the vaccine virus in stool samples was assessed by polymerase chain reaction (PCR).
  This endpoint was pre-specified to be analyzed in participants with IPV vaccination history.
Time Frame: Days 3, 5, 8, 10, 15, 22, 29, 36, 43, 50, and 57
Population: Participants in the Safety Population with available PCR data at each time point. The analysis includes groups with prior IPV history who received vaccination with a type 1 OPV.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History)
Number analyzed (Participants) | 18 | 18
percentage of participants
  Day 3: number analyzed (Participants) | 16 | 17
  Day 3 | 62.5 [35.4 to 84.8] | 82.4 [56.6 to 96.2]
  Day 5: number analyzed (Participants) | 15 | 13
  Day 5 | 93.3 [68.1 to 99.8] | 100 [75.3 to 100]
  Day 8: number analyzed (Participants) | 17 | 18
  Day 8 | 100 [80.5 to 100] | 100 [81.5 to 100]
  Day 10: number analyzed (Participants) | 17 | 16
  Day 10 | 100 [80.5 to 100] | 100 [79.4 to 100]
  Day 15: number analyzed (Participants) | 17 | 16
  Day 15 | 94.1 [71.3 to 99.9] | 81.3 [54.4 to 96.0]
  Day 22: number analyzed (Participants) | 18 | 16
  Day 22 | 50.0 [26.0 to 74.0] | 43.8 [19.8 to 70.1]
  Day 29: number analyzed (Participants) | 18 | 15
  Day 29 | 22.2 [6.4 to 47.6] | 26.7 [7.8 to 55.1]
  Day 36: number analyzed (Participants) | 13 | 15
  Day 36 | 30.8 [9.1 to 61.4] | 13.3 [1.7 to 40.5]
  Day 43: number analyzed (Participants) | 15 | 15
  Day 43 | 0.0 [0.0 to 21.8] | 6.7 [0.2 to 31.9]
  Day 50: number analyzed (Participants) | 18 | 14
  Day 50 | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 23.2]
  Day 57: number analyzed (Participants) | 16 | 14
  Day 57 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 23.2]
  At any time point | 100 [81.5 to 100] | 100 [81.5 to 100]

20. Secondary Outcome: Percentage of Participants Shedding Type 3 Vaccine Virus at Each Post-vaccination Stool Collection in Participants With IPV Vaccination History
Description: as for outcome 19
Time Frame: Days 3, 5, 8, 10, 15, 22, 29, 36, 43, 50, and 57
Population: Participants in the Safety Population with available PCR data at each time point. The analysis includes groups with prior IPV history who received vaccination with a type 3 OPV
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History)
Number analyzed (Participants) | 19 | 15
percentage of participants
  Day 3: number analyzed (Participants) | 17 | 14
  Day 3 | 88.2 [63.6 to 98.5] | 71.4 [41.9 to 91.6]
  Day 5: number analyzed (Participants) | 17 | 12
  Day 5 | 100 [80.5 to 100] | 100 [73.5 to 100]
  Day 8: number analyzed (Participants) | 17 | 14
  Day 8 | 100 [80.5 to 100] | 100 [76.8 to 100]
  Day 10: number analyzed (Participants) | 16 | 13
  Day 10 | 93.8 [69.8 to 99.8] | 100 [75.3 to 100]
  Day 15: number analyzed (Participants) | 17 | 15
  Day 15 | 76.5 [50.1 to 93.2] | 93.3 [68.1 to 99.8]
  Day 22: number analyzed (Participants) | 18 | 13
  Day 22 | 38.9 [17.3 to 64.3] | 61.5 [31.6 to 86.1]
  Day 29: number analyzed (Participants) | 18 | 14
  Day 29 | 38.9 [17.3 to 64.3] | 50.0 [23.0 to 77.0]
  Day 36: number analyzed (Participants) | 18 | 12
  Day 36 | 27.8 [9.7 to 53.5] | 33.3 [9.9 to 65.1]
  Day 43: number analyzed (Participants) | 17 | 14
  Day 43 | 11.8 [1.5 to 36.4] | 7.1 [0.2 to 33.9]
  Day 50: number analyzed (Participants) | 17 | 14
  Day 50 | 0.0 [0.0 to 19.5] | 7.1 [0.2 to 33.9]
  Day 57: number analyzed (Participants) | 17 | 15
  Day 57 | 0.0 [0.0 to 19.5] | 6.7 [0.2 to 31.9]
  At any time point | 100 [82.4 to 100] | 100 [78.2 to 100]

21. Secondary Outcome: Amount of Type 1 Vaccine Virus in Each Stool Sample Positive for Virus in Participants With IPV Vaccination History
Description: Samples positive for vaccine virus in stool as detected by PCR were quantified using a cell culture infectious dose assay. Participants who were PCR-positive for type 1 viral shedding but with log₁₀ CCID50 per gram ≤ LLOQ contributed a value equal to the LLOQ.
  This endpoint was pre-specified to be analyzed in participants with IPV vaccination history.
Time Frame: Days 3, 5, 8, 10, 15, 22, 29, 36, 43, 50, and 57
Population: Participants in the Safety population who were PCR-positive for poliovirus type 1 viral shedding and with available CCID50 data. The analysis includes groups with prior IPV history who received vaccination with a type 1 OPV.
Measure: Median (95% Confidence Interval); unit: log₁₀ CCID50 per gram
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History)
Number analyzed (Participants) | 18 | 18
log₁₀ CCID50 per gram
  Day 3: number analyzed (Participants) | 10 | 14
  Day 3 | 2.94 [2.750 to 3.875] | 3.22 [2.750 to 4.211]
  Day 5: number analyzed (Participants) | 14 | 13
  Day 5 | 3.22 [2.922 to 4.125] | 4.28 [3.906 to 4.875]
  Day 8: number analyzed (Participants) | 17 | 18
  Day 8 | 3.41 [2.813 to 4.000] | 4.33 [4.109 to 4.609]
  Day 10: number analyzed (Participants) | 17 | 16
  Day 10 | 3.19 [2.938 to 3.719] | 4.08 [3.063 to 4.531]
  Day 15: number analyzed (Participants) | 16 | 13
  Day 15 | 2.75 [2.750 to 2.813] | 2.75 [2.750 to 2.781]
  Day 22: number analyzed (Participants) | 9 | 7
  Day 22 | 2.75 [2.750 to 3.219] | 2.75 [2.750 to 3.313]
  Day 29: number analyzed (Participants) | 4 | 4
  Day 29 | 2.77 [2.750 to 2.781] | 2.88 [2.750 to 3.625]
  Day 36: number analyzed (Participants) | 4 | 2
  Day 36 | 2.75 [2.750 to 3.313] | 2.91 [2.750 to 3.063]
  Day 43: number analyzed (Participants) | 0 | 1
  Day 43 |  | 3.34 [3.34 to 3.34]
  Day 50: number analyzed (Participants) | 0 | 0
  Day 57: number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Amount of Type 3 Vaccine Virus in Each Stool Sample Positive for Virus in Participants With IPV Vaccination History
Description: Samples positive for vaccine virus in stool as detected by PCR were quantified using a cell culture infectious dose assay. Participants who were PCR-positive for type 3 viral shedding but with log₁₀ CCID50 per gram ≤ LLOQ contributed a value equal to the LLOQ.
  This endpoint was pre-specified to be analyzed in participants with IPV vaccination history.
Time Frame: Days 3, 5, 8, 10, 15, 22, 29, 36, 43, 50, and 57
Population: Participants in the Safety population who were PCR-positive for poliovirus type 3 viral shedding. The analysis includes groups with prior IPV history who received vaccination with a type 3 OPV.
Measure: Median (95% Confidence Interval); unit: log₁₀ CCID50 per gram
Arm/Group | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History)
Number analyzed (Participants) | 19 | 15
log₁₀ CCID50 per gram
  Day 3: number analyzed (Participants) | 15 | 10
  Day 3 | 4.06 [2.938 to 4.750] | 4.00 [2.781 to 4.734]
  Day 5: number analyzed (Participants) | 17 | 12
  Day 5 | 3.88 [2.906 to 4.500] | 4.23 [3.063 to 4.672]
  Day 8: number analyzed (Participants) | 17 | 14
  Day 8 | 4.28 [3.094 to 4.594] | 4.42 [3.094 to 4.875]
  Day 10: number analyzed (Participants) | 15 | 13
  Day 10 | 4.16 [2.844 to 4.375] | 3.97 [3.000 to 4.938]
  Day 15: number analyzed (Participants) | 13 | 14
  Day 15 | 2.84 [2.750 to 3.063] | 3.02 [2.766 to 3.469]
  Day 22: number analyzed (Participants) | 7 | 8
  Day 22 | 2.75 [2.750 to 2.781] | 3.09 [2.875 to 4.125]
  Day 29: number analyzed (Participants) | 7 | 7
  Day 29 | 2.75 [2.750 to 2.813] | 2.78 [2.750 to 2.844]
  Day 36: number analyzed (Participants) | 5 | 4
  Day 36 | 2.78 [2.750 to 3.281] | 2.75 [2.750 to 3.844]
  Day 43: number analyzed (Participants) | 2 | 1
  Day 43 | 2.77 [2.750 to 2.781] | 2.97 [2.97 to 2.97]
  Day 50: number analyzed (Participants) | 0 | 1
  Day 50 |  | 2.81 [2.81 to 2.81]
  Day 57: number analyzed (Participants) | 0 | 1
  Day 57 |  | 3.78 [3.78 to 3.78]

23. Secondary Outcome: Shedding Index of Vaccine Virus Shedding in Stool in Participants With IPV Vaccination History
Description: The Shedding Index Endpoint (SIE) was computed as the mean of the log₁₀ cell culture infectious dose 50% (CCID50) per gram from nominal collection days 7, 14, 21, and 28 post-dose (i.e., study days 8, 15, 22, and 29). Participants who were PCR-positive for type-specific viral shedding but with log₁₀ CCID50 per gram ≤ LLOQ contributed a value equal to the LLOQ.
  This endpoint was pre-specified to be analyzed in participants with IPV vaccination history.
Time Frame: Days 8, 15, 22, and 29
Population: Participants with complete data at all four time points (Days 8, 15, 22, and 29) were included in the analysis. The analysis includes groups with prior IPV history.
Measure: Median (95% Confidence Interval); unit: log₁₀ CCID50 per gram
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History) | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History)
Number analyzed (Participants) | 16 | 13 | 14 | 11
log₁₀ CCID50 per gram | 1.88 [1.477 to 2.344] | 1.96 [1.734 to 2.477] | 2.20 [1.844 to 3.016] | 2.41 [1.766 to 3.578]

24. Secondary Outcome: Area Under the Curve From Vaccination to 28 Days After Vaccination (AUC₀-₂₈) of Vaccine Virus Shed in Stool in Participants With an IPV Vaccination History
Description: Area under the curve (AUC) was computed for each participant using CCID50 per gram data collected through Day 29 using the linear trapezoidal rule. Participants were assumed to be not shedding at time of vaccination (i.e. there was no stool collection on Day 1). Participants who were PCR-positive for type-specific viral shedding but with log₁₀ CCID50 per gram ≤ LLOQ contributed a value equal to the LLOQ.
  This endpoint was pre-specified to be analyzed in participants with IPV vaccination history.
Time Frame: Days 3, 5, 8, 10, 15, 22, and 29
Population: Participants with available CCID50/g shedding data (must have data from Day 3 and Day 29, and no 2 missing consecutive samples from Days 5, 8, 10, 15, and 22). The analysis includes groups with prior IPV history.
Measure: Median (95% Confidence Interval); unit: days * log₁₀ CCID50/gram
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History) | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History)
Number analyzed (Participants) | 15 | 15 | 17 | 12
days * log₁₀ CCID50/gram | 57.84 [10.188 to 66.625] | 66.88 [52.797 to 78.344] | 60.80 [49.172 to 80.438] | 71.46 [56.711 to 87.945]

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious AEs were collected up to Day 169. Non-serious AEs were collected up to 28 days after each vaccination (Day 1-28 for 1st vaccination and Day 29-56 for the 2nd vaccination). Solicited AEs were collected up to 7 days after each vaccination (Days 1-7 for 1st vaccination and Days 29-35 for the 2nd vaccination).
Description: All-cause mortality is reported for all randomized participants. AEs are reported for the Reactogenicity Population, defined as all participants who provided informed consent and received a study vaccine.
Arm/Group | Group1: nOPV1 (IPV History) | Group 2: mOPV1 (IPV History) | Group 3: nOPV1 (OPV History) | Group 4: mOPV1 (OPV History) | Group 5: nOPV3 (IPV History) | Group 6: mOPV3 (IPV History) | Group 7: nOPV3 (OPV History) | Group 8: mOPV3 (OPV History)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23 | 0/53 | 0/27 | 0/20 | 0/21 | 0/40 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/50 | 0/25 | 0/19 | 0/17 | 0/35 | 0/19
Other Adverse Events (participants affected / at risk) | 13/20 | 13/20 | 39/50 | 21/25 | 12/19 | 10/17 | 15/35 | 12/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group1: nOPV1 (IPV History) (N=20) | Group 2: mOPV1 (IPV History) (N=20) | Group 3: nOPV1 (OPV History) (N=50) | Group 4: mOPV1 (OPV History) (N=25) | Group 5: nOPV3 (IPV History) (N=19) | Group 6: mOPV3 (IPV History) (N=17) | Group 7: nOPV3 (OPV History) (N=35) | Group 8: mOPV3 (OPV History) (N=19)
Fatigue (General disorders) | 5 | 8 | 21 | 11 | 7 | 8 | 9 | 7
Chills (General disorders) | 1 | 5 | 3 | 3 | 1 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 11 | 10 | 3 | 7 | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 7 | 4 | 6 | 1 | 5 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 8 | 3 | 1 | 1 | 8 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 7 | 16 | 10 | 3 | 6 | 8 | 5
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 6 | 10 | 6 | 2 | 2 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4 | 6 | 1 | 2 | 2 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 2 | 2 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 2 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Immunisation reaction (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wisdom teeth removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsilitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that there should be a joint publication first; after the joint publication or after 24 months without a joint publication from the time of last participant last visit, the PI has a right to present the trial results at meetings or do their own publication in a journal, but they must provide PATH the chance to review the manuscript 60 days in advance of publication.

DOCUMENTS (2):
  • Study Protocol (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT04529538/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT04529538/SAP_001.pdf